CLINICAL TRIAL: NCT05924464
Title: Group Preconception Care for Fertility Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pomelo Care, Inc. (Unknown); Independence Blue Cross (Other)
Responsible Party: Principal Investigator, Anuja Dokras, Director of the Penn PCOS Center, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 852900
Record Dates: First submitted 2023-05-26; First posted 2023-06-29 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Group preconception care
  Interventions: Other: Group Preconception Care
- Control arm (No Intervention): Usual care (completion of questionnaires only)

INTERVENTIONS:
Other: Group Preconception Care — Groups of 6-10 patients to initiate biweekly virtual group care sessions on a rolling basis, with completion of enrollment and the virtual curriculum within a year.
  Arms: Intervention arm

SUMMARY:
Group Preconception Care for Fertility Patients aims to translate the well-established group prenatal care model to preconception care to improve pregnancy and neonatal outcomes. In partnership with Pomelo Care (a virtual maternity care program), the investigators are conducting this study using couples at Penn Fertility Care.

ELIGIBILITY:
Inclusion Criteria:

1. Female new patient seen at Penn Fertility Care for infertility or procreative management
2. Currently planning to conceive
3. Intending to carry pregnancy (i.e. will not need a gestational carrier), since our project aims to implement lifestyle changes prior to conception
4. Willing to be randomized to group preconception care versus usual care

Exclusion Criteria:

1. Prior infertility treatment at other practice in this initial project, we aim to focus on patients with a new diagnosis of infertility to allow time for completion of the virtual program during the diagnostic phase and early treatment phase
2. Known need for gestational carrier, as above
3. Planning preimplantation genetic testing for monogenic disorders or egg/embryo banking
4. Non-English speaking
5. Unable to complete electronic questionnaires due to lack of access to technology

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Blood pressure measurement recorded by clinician in Penn EMR | From enrollment to 16 weeks
  Was a blood pressure measurement recorded by a clinician in Penn EMR, yes/no
Weight measurement recorded by clinician in Penn EMR | From enrollment to 16 weeks
  Was a weight measurement recorded by a clinician in Penn EMR, yes/no
Hemoglobin A1c testing results recorded in Penn EMR | From enrollment to 16 weeks
  Was a hemoglobin A1c test performed if medically indicated (history of diabetes, BMI>30) or felt necessary by health care provider, yes/no
Change in Anxiety screening score | Enrollment, 4 months, 12 months
  Generalized Anxiety Disorder 7 (GAD-7) Questionnaire will be administered to both groups at enrollment, 4 months, and 12 months. The total score for the seven items ranges from 0 to 21, with 21 indicating a worse outcome
Change in Depression screening score | Enrollment, 4 months, 12 months
  Patient Health Questionnaire 9 (PHQ-9) will be administered to both groups at enrollment, 4 months, and 12 months. The total score for the nine items ranges from 0 to 27 where a high score indicates a worse outcome
Change in Fertility-related quality of life questionnaire score | Enrollment, 4 months, 12 months
  Fertility Related Quality of Life (FertiQOL) Questionnaire will be administered to both groups at enrollment, 4 months, and 12 months. The 36 FertiQoL items are rated according to 5 types of response scales. The total score is 100, with higher scores indicating worse fertility-related quality of life.
Incidence of ovulation stimulations | From enrollment to 12 months
  Count of ovarian stimulation treatments
Incidence of intrauterine inseminations | From enrollment to 12 months
  Count of intrauterine insemination treatments
Incidence of in vitro fertilizations | From enrollment to 12 months
  Count of in vitro fertilization treatments
Pregnancy rate | From enrollment to 12 months
  This includes the number of patients who become pregnant during the study period in both groups.
Time to pregnancy in days | From enrollment to 12 months
  This includes the time until patients become pregnant during the study period in both groups.
Patient experience | Enrollment to 16 weeks
  In the intervention arm only, brief questionnaires will be distributed after each virtual session to ask participants to rate their satisfaction with the session. Patients will also complete a cumulative evaluation at the conclusion of the sessions. These surveys will use a Likert scale with a higher score indicating a better experience.
Miscarriage rate | From enrollment up to 18 months
  Total number of miscarriages per participants who become pregnant in either group
Number of pregnant participants with occurrence of a hypertensive disorder of pregnancy | Conception to delivery, approximately 9 months
  This will be scored yes if any of the following are noted in the medical record: gestational hypertension (blood pressure >140/90 on 2 or more occasions at least 4 hours apart), severe preeclampsia (blood pressure >160/110 on 2 or more occasions at least 4 hours apart, or mildly elevated blood pressures with persistent headache, scotomata, platelet count <100,000/uL, liver function tests twice the upper limit of normal, or creatinine >1.1 mg/dL), HELLP syndrome (hemolysis, elevated liver enzymes, and low platelet count), or eclampsia (elevated blood pressure with seizures).
Number of pregnant participants with a diagnosis of gestational diabetes | Conception to delivery, approximately 9 months
  This will be scored yes if gestational diabletes is diagnosed. Gestational diabetes is diagnosed based on an abnormal 3-hour glucose tolerance test (1-hour test blood glucose >135mg/dL will be followed by a 3-hour test). Two or more abnormal values on the 3-hour test is diagnostic of gestational diabetes. Cutoffs are 95 fasting, 180 at 1 hour, 155 at 2 hours, and 140 at 3 hours.
Number of pregnant participants with occurrences with an antepartum hospitalizations | Conception to delivery, approximately 9 months
  This includes hospital admissions during the pregnancy for any pregnancy or non-pregnancy related complications.
Number of pregnant participants with preterm birth | At time of delivery
  Preterm delivery is defined as delivery at less than 37 weeks gestational age.
Number of pregnant participants with a cesarean delivery | At time of delivery
  In participants who become pregnant, the incidence of cesarean delivery
Number of pregnant participants with a NICU admission | From date of delivery to date of discharge from hospital postpartum, up to 6 weeks from delivery
  Infant admission to neonatal intensive care unit.
Number of PEC (Perinatal Evaluation Center)/emergency room visits in pregnant participants | From date of conception to delivery date, approximately 9 months
  Total number of any presentation to the Perinatal Evaluation Center or emergency room during pregnancy
Among those patients that become pregnant, delivery length of stay | From date of delivery to date of discharge from hospital postpartum, up to six weeks from delivery
  Length of stay from birth to discharge, measured in hours
Among those patients that become pregnant, score on the Edinburgh Postnatal Depression Scale | Between 2 to 6 weeks after delivery
  Edinburgh Postnatal Depression Scale will either be abstracted from the medical record, or if not administered clinically, will be administered by the study team. The total score for the ten items ranges from 0 to 30 with a higher score indicating a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Reproductive Research Unit, 3701 Market Street, Suite 810, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided